CLINICAL TRIAL: NCT06797882
Title: The Effectiveness of Silver Diamine Fluoride (SDF) in the Prevention of Early Enamel Caries Among Patients With Fixed Orthodontic Appliances: A Randomised Controlled Trial
Brief Title: Preventive Effects of Silver Diamine Fluoride on Early Enamel Caries
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Ahmad Shuhud Irfani bin Zakaria, Principal Investigator, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JEP-2024-878
Record Dates: First submitted 2025-01-27; First posted 2025-01-29 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Demineralization, Tooth; White Spot Lesion of Tooth; Fixed Appliances; Early Caries Lesions
Keywords: Early Caries Lesions; Silver Diamine Fluoride (SDF); Fixed Orthodontic Appliances; Caries Prevention; Fluoride Varnish; White Spot Lesions
MeSH Terms: conditions — Tooth Demineralization | interventions — silver diamine fluoride; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study follows a randomized controlled trial design with three parallel groups. Each participant, rather than specific areas within the mouth, will be the unit of randomization. This method, in contrast to a split-mouth design, helps prevent issues related to cross-contamination.
Who Masked: Participant, Outcomes Assessor
Masking Description: A total of 99 eligible participants will be randomly assigned to three intervention groups-SDF, FV (gold standard), or normal saline (placebo)-with 33 participants per group. Randomization will be conducted using Microsoft Excel by a data manager, who is not blinded and will ensure proper group allocation. Participants will be blinded to their assigned intervention, which will be provided in a concealed opaque envelope. The care provider, however, will not be blinded due to the distinct characteristics of each material. Follow-up assessments will occur at 1, 3, 6, and 12 months. At each visit, a blinded outcome assessor will evaluate the upper incisors using the ICDAS II scoring system and DIAGNOdent after prophylactic cleaning. Additionally, digital photographs will be assessed using the Gorelick scoring system by blinded outcome assessors on a separate occasion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of care + Silver Diamine Fluoride (SDF) (Experimental): Intervention 1 will receive standard OHI (every three months) and application of Silver Diamine Fluoride (SDF (Riva Star, SDI Limited., Australia) every six months.
  Interventions: Drug: Silver diamine fluoride- potassium iodide
- Standard of care + Fluoride varnish (Active Comparator): Intervention 2 will receive standard OHI (every three months) and application of topical fluoride varnish containing 5% NaF (Duraphat varnish®, Colgate-Palmolive (UK) Ltd) every six months.
  Interventions: Drug: Fluoride varnish
- Standard of care + Normal Saline (Placebo Comparator): Control will receive standard oral hygiene instructions (OHI every three months) and application of normal saline every six months.
  Interventions: Other: 0.9 % saline

INTERVENTIONS:
Drug: Silver diamine fluoride- potassium iodide — SDF , Riva Star, SDI Limited., Australia
  Other Names: Silver Diamine Fluoride
  Arms: Standard of care + Silver Diamine Fluoride (SDF)
Drug: Fluoride varnish — Duraphat varnish®, Colgate-Palmolive (UK) Ltd.
  Arms: Standard of care + Fluoride varnish
Other: 0.9 % saline — Standard oral hygiene instructions every 3 months and application of Normal Saline for every 6 months
  Arms: Standard of care + Normal Saline

SUMMARY:
Fixed orthodontic patients are at risk of developing dental caries. Topical application of fluoride varnish (FV) around the orthodontic brackets and using fluoridated mouth rinses have been suggested to prevent the formation of white spot lesions (WSLs) on enamel. Recent studies have shown that silver diamine fluoride (SDF) demonstrated better outcomes in dental caries prevention as compared to FV. However, the caries preventive effects of SDF application around the orthodontic brackets have not been established yet.

This study will be conducted to evaluate the effectiveness of SDF in preventing WSLs formation in patients undergoing fixed orthodontic treatment. This study will use a randomised-controlled double-blinded design with three parallel arms. Ninety-nine eligible participants will be recruited. Using their registration number, a random list of patients will be generated using computer software. Each patient will be assigned randomly to three groups: SDF, FV, or placebo. Digital photographs of upper anterior teeth (frontal view) will be taken as a baseline and repeated at every review appointment. The materials will be applied around the orthodontic bracket of upper incisors and canines every 6 months. The formation of WSLs around the bracket will be evaluated at 1, 3, 6, and 12 months using three parameters: the ICDAS scoring system, the laser fluorescence caries detector, and digital photographic analysis using the Gorelick score. The patients' perception of the colour changes of the enamel will be evaluated through patient-reported outcomes. The difference in ICDAS and Gorelick scores and the patients' perceptions will be reported through descriptive statistics. The Kruskal-Wallis or one-way ANOVA statistical test will be used to compare the changes in fluorescence intensity between treatment groups.

The investigators believe that the results of this study will provide insight into the caries preventive protocol among fixed orthodontics patients and subsequently reduce the incidence of WSLs during orthodontic treatment.

DETAILED DESCRIPTION:
Fixed orthodontic appliances are commonly used to correct malocclusions and align teeth in orthodontic treatment. Fixed orthodontic appliances consist of several components, each serving a specific function in the orthodontic treatment process. These components typically include brackets, arch wires, ligatures (or ties), and occasionally auxiliary components such as springs or elastics. It involves the placement of orthodontic brackets, secured to the teeth surface with a composite resin material. Slots on the brackets are used to hold the orthodontic wires, which act as a means of transmitting forces to the teeth for their movement during orthodontic treatment.

The direct bonding of orthodontic devices to teeth has had a profound impact on orthodontic practices. In the early days of orthodontic treatment, brackets were attached to gold or stainless-steel bands. This process was time-consuming and uncomfortable for patients, often causing gingival trauma and decalcification. In the mid-1960s, researchers pioneered the bonding of brackets directly to enamel. Since then, there have been numerous advancements in adhesives, base designs, bracket materials, curing methods, primers, fluoride-releasing agents, and sealants. Nevertheless, the incidence and severity of white spot lesions caused by enamel decalcification are increasing among those receiving orthodontic treatment. Surprisingly, these lesions can appear as early as one month after the placement of orthodontic brackets. Prolonged treatment, lasting over a year, increases this risk due to the presence of fixed appliances, creating areas for plaque accumulation. This plaque may rapidly modify the composition of bacteria, particularly acid-producing bacteria, leading to enamel erosion and the formation of white spot lesions (WSLs).

White spot lesions are rapidly forming, prompting clinicians to explore solutions for orthodontic-associated demineralization. Factors such as food debris, diet, fluoride availability, mineral crystal composition, and salivary content can influence demineralization periods. Studies have shown that preventive strategies, such as application of topical fluorides, reduce the incidence of WSLs formation. A systematic review has demonstrated the effectiveness of topical sodium fluoride varnishes (FV) in preventing enamel decalcification during orthodontic treatment with fixed appliances. However, the reported preventive fraction is wide, ranging from 12 to 55%. This shows that the preventive effects of FV are not consistent and vary between individuals. The range of results seen may also be attributed to the bioavailability of fluoride in saliva, which is regulated by variables including salivary secretion rate, dietary fluoride consumption, and the usage of fluoridated products. While traditional fluorides like sodium fluoride support remineralization following topical application, they exhibit shorter persistence in saliva compared to SDF's 38% retention. This is due to the stable silver halide compound that forms in saliva, which helps sustain SDF over an extended period of time, and the high fluoride content of SDF, which renders it a great potential for remineralization. Further, the remineralisation and antibacterial effects of fluoride are slow and highly dependent on factors such as patients brushing efficacy and the stability of the fluoride ion in the saliva. This might explain why the WSLs are still occur and present around the orthodontic brackets even though the preventive measures have been implemented.

Recently, the use of silver diamine fluoride (SDF) has gained much attention in caries management strategy, especially on cavitated lesions. SDF was introduced into the dental field by Nishiino, Yamaga and their colleagues in the 1960s available at 38% concentration. SDF is a colourless and odorless solution which consists of silver, fluoride, and ammonia ion. The presence of the silver component in the SDF formulation helps in stimulating dentine sclerosis and provides antibacterial activity by causing immediate bacterial death through inhibition of bacterial DNA replication and blocking the formation of proteolytic enzymes. Fluoride on the other hand act as a remineralising agent and presents at a high concentration of 44,800 ppm.

The combined effects of remineralising and antibacterial properties make SDF an effective cariostatic agent. A systematic review showed that SDF effectively arrests decay in primary teeth in children, with a proportion of 66%-81% with annual or biannual application, while it was reported that the preventive fraction of SDF is as high as 61% and 72%, respectively. In comparison to fluoride varnish, SDF has a better caries arrest ability on both primary and permanent teeth, where the effectiveness is almost doubled than the effects of sodium fluoride varnish at 30 months.

The only drawback of SDF application is the formation of black staining on the cavitated lesion due to the formation of silver phosphate precipitate when hydroxyapatite crystals react with the SDF solution. However, the addition of potassium iodide managed to reduce the staining effects, leading to a yellow-brown rather than a black discoloration. In addition, SDF will not stain sound enamel suggesting its promising role in the prevention of dental caries.

However, based on our knowledge, the effects of SDF in preventing WSLs formation in patients with fixed orthodontics has not been established yet. Therefore, the investigators would like to take this opportunity and conduct a clinical trial with the aim to investigate the effectiveness of Silver Diamine Fluoride (SDF) in caries prevention among patients with fixed orthodontic appliances.

ELIGIBILITY:
Inclusion Criteria:

* Subjects about to undergo fixed orthodontic treatment at the Faculty of Dentistry, UKM.
* Subjects must be aged 18 years and above.
* Consented for treatment. Patients will be informed of the risk and benefit of the study for each treatment group through the patient information sheet given to them before obtaining their consent.
* Orthodontic brackets placed at least on the upper incisors.
* Patients undergoing orthodontic treatment with conventional orthodontic brackets placed on the labial surface.
* Any degree of malocclusion
* Fit and healthy patient
* Non-smoker
* Subjects can understand and possessed basic command in English

Exclusion Criteria:

* History of fixed orthodontic treatment
* Presence of any dental anomalies or developmental defects of enamel (DDE) on labial surfaces of teeth, such as preexisting fluorosis or enamel hypoplasia.
* Presence of any or direct/indirect restorations on the labial surface of teeth
* History of long-term antibiotic usage
* Presence of untreated cavitated lesions, especially on upper and lower incisors and canines
* Plaque levels >30%.
* Patient allergic to any of the content of the intervention material (sodium fluoride, silver diamine fluoride, potassium iodide).
* Patients with lingual brackets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Formation of Early Enamel Caries Analyzed Through Digital Photography | 12 months
  Changes in enamel surface following decalcification, measured using the Gorelick's Index (1982) in all three intervention groups.
  Gorelick's Index Scale:
  0 - No lesion (best outcome)
  1. - Moderate lesion
  2. - Severe lesion
  3. - Cavitation (worst outcome) Lower scores represent better outcomes, while higher scores indicate poorer outcomes.
Formation of Early Enamel Caries Assessed Clinically by a Blinded Assessor | 12 months
  Changes in enamel surface following decalcification, measured clinically using the International Caries Detection and Assessment System II (ICDAS II) Index (2005) in all three intervention groups.
  ICDAS II Scale:
  0 - Sound tooth surface: No evidence of caries after 5 seconds of air drying (best outcome)
  1. - First visual change in enamel: Opacity or discoloration (white or brown) visible after prolonged air drying
  2. - Distinct visual change in enamel visible when wet; lesion must be visible when dry
  3. - Localized enamel breakdown (without clinical visual signs of dentinal involvement), seen when wet and after prolonged drying
  4. - Underlying dark shadow from dentine
  5. - Distinct cavity with visible dentine
  6. - Extensive (more than half the surface) distinct cavity with visible dentine (worst outcome) Lower scores represent better outcomes, while higher scores indicate poorer outcomes.
Change in Laser Fluorescence Values | 12 months
  Changes in mean DIAGNOdent scores among the three study groups.
  DIAGNOdent Scale:
  0-13 - Sound tooth surface (best outcome) 14-20 - Enamel caries >20 - Dentinal caries (worst outcome) Lower readings represent better outcomes, while higher readings indicate poorer outcomes.
Participants Perspectives on Tooth Colour Changes After Silver Diamine Fluoride (SDF) Application: Participants-Reported Outcome | 12 months
  Participants perceptions of visible colour changes following SDF application will be evaluated using a structured questionnaire at baseline and follow-up appointments (1, 3, 6, and 12 months). Participants will report whether they notice any colour changes and indicate their satisfaction with the appearance of their teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Shuhud Irfani Zakaria, MClinDent, Principal Investigator — National University of Malaysia
Locations (1):
- Faculty of Dentistry, UKM, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
Data will be submitted to the university repository and final data will be deposited to the university. Patient personal information will be protected and subjected to Data Security Act.

REFERENCES:
- [Background] Mungur A, Chen H, Shahid S, Baysan A. A systematic review on the effect of silver diamine fluoride for management of dental caries in permanent teeth. Clin Exp Dent Res. 2023 Apr;9(2):375-387. doi: 10.1002/cre2.716. Epub 2023 Feb 23. PMID 36823765
- [Background] Lussi A, Megert B, Longbottom C, Reich E, Francescut P. Clinical performance of a laser fluorescence device for detection of occlusal caries lesions. Eur J Oral Sci. 2001 Feb;109(1):14-9. doi: 10.1034/j.1600-0722.2001.109001014.x. PMID 11330928
- [Background] Lazar L, Vlasa A, Beresescu L, Bud A, Lazar AP, Matei L, Bud E. White Spot Lesions (WSLs)-Post-Orthodontic Occurrence, Management and Treatment Alternatives: A Narrative Review. J Clin Med. 2023 Feb 28;12(5):1908. doi: 10.3390/jcm12051908. PMID 36902696
- [Background] Jabin Z, Nasim I, Priya V V, Agarwal N. Comparative Evaluation of Salivary Fluoride Concentration after Topical Application of Silver Diamine Fluoride and Sodium Fluoride: A Randomized Controlled Trial. Int J Clin Pediatr Dent. 2022 May-Jun;15(3):371-375. doi: 10.5005/jp-journals-10005-2398. PMID 35991787
- [Background] Hicks J, Garcia-Godoy F, Flaitz C. Biological factors in dental caries: role of remineralization and fluoride in the dynamic process of demineralization and remineralization (part 3). J Clin Pediatr Dent. 2004 Spring;28(3):203-14. doi: 10.17796/jcpd.28.3.w0610427l746j34n. PMID 15163148
- [Background] Gange P. The evolution of bonding in orthodontics. Am J Orthod Dentofacial Orthop. 2015 Apr;147(4 Suppl):S56-63. doi: 10.1016/j.ajodo.2015.01.011. PMID 25836345
- [Background] Seifo N, Robertson M, MacLean J, Blain K, Grosse S, Milne R, Seeballuck C, Innes N. The use of silver diamine fluoride (SDF) in dental practice. Br Dent J. 2020 Jan;228(2):75-81. doi: 10.1038/s41415-020-1203-9. PMID 31980777
- [Background] Tufekci E, Dixon JS, Gunsolley JC, Lindauer SJ. Prevalence of white spot lesions during orthodontic treatment with fixed appliances. Angle Orthod. 2011 Mar;81(2):206-10. doi: 10.2319/051710-262.1. PMID 21208070
- [Background] Sonesson M, Twetman S. Prevention of white spot lesions with fluoride varnish during orthodontic treatment with fixed appliances: a systematic review. Eur J Orthod. 2023 Sep 18;45(5):485-490. doi: 10.1093/ejo/cjad013. PMID 37032523
- [Background] Sardana D, Ekambaram M, Yang Y, McGrath CP, Yiu CKY. Caries-preventive effectiveness of two different fluoride varnishes: A randomised clinical trial in patients with multi-bracketed fixed orthodontic appliances. Int J Paediatr Dent. 2023 Jan;33(1):50-62. doi: 10.1111/ipd.13013. Epub 2022 Jul 10. PMID 35737872
- [Background] Sardana D, Li KY, Ekambaram M, Yang Y, McGrath CP, Yiu CK. Validation of clinical photography and a laser fluorescence device for assessment of enamel demineralization during multi-bracketed fixed orthodontic treatment. Photodiagnosis Photodyn Ther. 2022 Jun;38:102828. doi: 10.1016/j.pdpdt.2022.102828. Epub 2022 Mar 23. PMID 35339722
- [Background] Kidd E, Fejerskov O. Changing concepts in cariology: forty years on. Dent Update. 2013 May;40(4):277-8, 280-2, 285-6. doi: 10.12968/denu.2013.40.4.277. PMID 23829008
- [Background] Jiang H, Hua F, Yao L, Tai B, Du M. Effect of 1.23% acidulated phosphate fluoride foam on white spot lesions in orthodontic patients: a randomized trial. Pediatr Dent. 2013 May-Jun;35(3):275-8. PMID 23756315
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Background] Horst JA, Heima M. Prevention of Dental Caries by Silver Diamine Fluoride. Compend Contin Educ Dent. 2019 Mar;40(3):158-163; quiz 164. PMID 30829497
- [Background] Gorelick L, Geiger AM, Gwinnett AJ. Incidence of white spot formation after bonding and banding. Am J Orthod. 1982 Feb;81(2):93-8. doi: 10.1016/0002-9416(82)90032-x. PMID 6758594
- [Background] Duangthip D, Fung MHT, Wong MCM, Chu CH, Lo ECM. Adverse Effects of Silver Diamine Fluoride Treatment among Preschool Children. J Dent Res. 2018 Apr;97(4):395-401. doi: 10.1177/0022034517746678. Epub 2017 Dec 13. PMID 29237131
- [Background] Chu CH, Lo EC, Lin HC. Effectiveness of silver diamine fluoride and sodium fluoride varnish in arresting dentin caries in Chinese pre-school children. J Dent Res. 2002 Nov;81(11):767-70. doi: 10.1177/0810767. PMID 12407092
- [Background] Camacho KJ, English JD, Jacob HB, Harris LM, Kasper FK, Bussa HI, Quock RL. Silver diamine fluoride and bond strength to enamel in vitro: A pilot study. Am J Dent. 2018 Dec;31(6):317-319. PMID 30658379
- [Background] Bishara SE, Gordan VV, VonWald L, Jakobsen JR. Shear bond strength of composite, glass ionomer, and acidic primer adhesive systems. Am J Orthod Dentofacial Orthop. 1999 Jan;115(1):24-8. doi: 10.1016/s0889-5406(99)70312-4. PMID 9878954
- [Background] Crystal YO, Janal MN, Hamilton DS, Niederman R. Parental perceptions and acceptance of silver diamine fluoride staining. J Am Dent Assoc. 2017 Jul;148(7):510-518.e4. doi: 10.1016/j.adaj.2017.03.013. Epub 2017 Apr 27. PMID 28457477